CLINICAL TRIAL: NCT06769035
Title: Effect of a Food Supplement with Extracts of Cocoa, Amaranth Seed and Ginger in Overweight or Obese Patients in the Outpatient Clinic of the New Juan I. Menchaca Civil Hospital
Brief Title: Effect of a Food Supplement with Natural Extracts of Cocoa, Amaranth Seed and Ginger in Overweight or Obese Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Luis Miguel Román Pintos, Doctor in pharmacology and internist. Professor at University of Guadalajara, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 00082
Record Dates: First submitted 2024-12-13; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Oxidative Stress; Inflammation Biomarkers; Obesity and Overweight
Keywords: Food supplement; Cocoa; Amaranth seed; Ginger; Oxidative stress; Inflammation
MeSH Terms: conditions — Obesity; Overweight; Inflammation | interventions — Chocolate; ginger extract

STUDY DESIGN:
Intervention Model Description: Clinical trial, randomized, double-blind, controlled with a placebo group, 40 patients between 18 and 60 years of age, with the presence of overweight, will be divided into parallel groups, group A cocoa, amaranth seed and ginger, group B cocoa, group C amaranth, group D placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Food supplement: cocoa, amaranth seed and ginger (Active Comparator): Group A:
  20g Cocoa, 10g amaranth seed and 1g ginger once a day for 12 weeks
  Interventions: Dietary Supplement: Cocoa, amaranth seed and ginger
- Food supplement: cocoa (Active Comparator): Group B:
  20g Cocoa once a day for 12 weeks
  Interventions: Dietary Supplement: Cocoa
- Food supplement: amaranth (Active Comparator): Group C:
  10g Amaranth seed once a day for 12 weeks
  Interventions: Dietary Supplement: Amaranth seed
- Food supplement: placebo (Placebo Comparator): Group D:
  Coloring and flavoring, one dose per day for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cocoa, amaranth seed and ginger — Sachet with 20gr of cocoa, 10g of amaranth seed and 1g of ginger, one dose per day for 12 weeks
  Other Names: cocoa; ginger; amaranth seed
  Arms: Food supplement: cocoa, amaranth seed and ginger
Dietary Supplement: Amaranth seed — Sachet with 10g of amaranth seed one dose per day for 12 weeks
  Arms: Food supplement: amaranth
Dietary Supplement: Cocoa — Sachet with 20gr of cocoa one dose per day for 12 weeks
  Arms: Food supplement: cocoa
Dietary Supplement: Placebo — Sachet with coloring and flavoring, one dose per day for 12 weeks one dose per day for 12 weeks
  Arms: Food supplement: placebo

SUMMARY:
Clinical trial, randomized, double-blind, controlled with a placebo group, 40 patients between 18 and 60 years of age, with the presence of overweight, will be divided into parallel groups, group A cocoa, amaranth seed and ginger, group B cocoa, group C amaranth, group D placebo, with the objective of evaluating the effect of the nutritional supplement in overweight or obese patients on cytokines, insulin resistance and oxidative stress. The study consists of 4 visits: screening (-21 days), baseline (day 0), follow-up (week 6) and end of the study (12 weeks) and 2 follow-up calls (weeks 3 and 10). For 12 weeks they will take one sachet of the supplement containing cocoa, amaranth seed and ginger or placebo daily. Waist circumference, somatometric parameters, vital signs, nocturnal decrease in blood pressure, ankle arm index, cytokines, glucose, glycated hemoglobin, hs-CRP, lipid profile, insulin, antioxidant effect, blood cytometry, function tests will be evaluated. liver, urea, creatinine, uric acid and urine pregnancy test for women of childbearing age. A 24-hour reminder and frequency of consumption will be carried out to assess the diet at each of the visits and nutritional recommendations will be given. Adherence to treatment (Morisky-Green), adverse events and concomitant treatments will be verified throughout the study.

DETAILED DESCRIPTION:
Overweight and obesity are a public health problem with worldwide prevalence and play an important role in the emergence of chronic diseases. Overweight is characterized by low-grade chronic inflammation and is associated with an abnormal inflammatory response, oxidative stress and low sensitivity. to insulin. Inflammation of adipose tissue is initiated and sustained over time by dysfunctional adipocytes that secrete inflammatory adipokines; elevated proinflammatory stimuli directly affect insulin signaling in target tissues. Oxidative stress alters mitochondrial activity, modifies the concentration of inflammation levels associated with many adipocytes, promotes lipogenesis, stimulates the change of preadipocytes for mature adipocytes and regulates the energy balance in neurons that control appetite. It is also an important regulator. of insulin sensitivity.

The solution to the consequences of obesity and overweight, low-grade inflammation, oxidative stress and insulin sensitivity are based on pharmaceutical treatments and surgical processes, but changes in lifestyle are the cornerstone of treatment, however the patient's adherence to treatment is low and the results are long-term, for this reason some authors have dedicated themselves to looking for alternatives that complement changes in lifestyle and improve health status.

Polyphenols are bioactive compounds that have been shown to influence insulin resistance, oxidative stress and inflammation. There is extensive evidence from clinical studies and meta-analyses in overweight patients to support the effects of this study's supplement on waist circumference, weight, BMI, blood pressure, insulin sensitivity, markers of inflammation, and oxidative stress.

Cocoa has been positioned as a preventive phytopharmaceutical due to its polyphenolic compounds, mainly flavonols with anti-inflammatory and antioxidant effects, which can help prevent or delay the complications of DM2 by modulating insulin secretion.

Amaranth seed is a source of protein, calcium, iron, dietary fiber, vitamin E and D, with a high content of monounsaturated fats and polyunsaturated fatty acids such as squalene, which have been given anti-inflammatory and antioxidant properties, Mozak and collaborators in 2018 did a clinical trial with amaranth seed in overweight patients with favorable results in reducing fasting insulin and the HOMA-IR index.

Ginger has been widely studied due to its potential in reducing glucose, lipid and body fat levels, and has been used as a preventative in chronic diseases. A clinical trial conducted in 2019 by Rahimlou and collaborators included 37 participants with metabolic syndrome, significantly decreased fasting glucose levels and improved insulin resistance.

The objective of the present study is to evaluate the effect of a supplement with cocoa, amaranth seed and ginger in overweight patients on inflammation, insulin resistance and oxidative stress.

ELIGIBILITY:
Inclusion criteria

1. Signed informed consent;
2. Men or women;
3. Age between 18 and 60 years;
4. Waist circumference ≥ 88 cm in women or ≥ 94 cm in men;
5. Plus one of the following criteria:

   * BMI >25 kg/m2 and not > 30 kg/m2 in both genders or history of bariatric surgery > 6 months;
   * Fasting serum glucose of 100-125 mg/dL or HbA1c of 5.7-6.4% or on pharmacological treatment with OAD for prediabetes;
   * Insulin resistance by HOMA > 2.6 and insulin sensitivity by QUICKI <0.34;F.
   * Negative pregnancy test.

Exclusion criteria

1. On pharmacological treatment or diet for weight control;
2. Routine use of antioxidants in the last 3 months;
3. BMI ≥ 30 kg/m2 or recent bariatric surgery (< 6 months);
4. LDL cholesterol > 160 mg/dL or total cholesterol > 200 mg/dL, and no treatment for dyslipidemia;
5. Major micro or macrovascular complications due to severe metabolic disease (history of acute coronary syndrome, cerebrovascular disease, peripheral arterial insufficiency or aortic aneurysm);
6. Pregnancy or breastfeeding;
7. Refusal to use an effective contraceptive method for the duration of the study;
8. Hypersensitivity to any of the components of the formula or phenylketonurics;
9. Endocrinological or rheumatic diseases;
10. Patient with recent initiation of vigorous physical exercise or exercise routine for weight loss and/or;
11. Liver or kidney failure by clinical and/or laboratory criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Insulin Resistance (IR) at 3 months | Change from baseline visit to final 3 months
  Average baseline and final HOMA-IR index
Change from baseline in oxidative stress markers Superoxide Dismutase (SOD), Catalase (CAT) and Glutathione Peroxidase (GPX) | Change from baseline visit to final 3 months
  Basal and final average of SOD, CAT and GPX

SECONDARY OUTCOMES:
Change in metabolic variables (Weight, kg) (Height, m) (Body Mass Index BMI) | Change from baseline visit to final 3-month period
  Average baseline and final visit (Weight, kg) (Height, m) in combination for BMI (Body Mass Index, kg/m2)
Change in metabolic variables (Waist Circumference WC, cm) | Change from baseline visit to final 3-month period
  Average baseline and final visit (Waist Circumference WC, cm)
Change in metabolic variables (% fat, % visceral fat) | Change from baseline visit to final 3-month period
  Average baseline and final visit (% fat, % visceral fat)
Change in metabolic variables (Muscle Mass MM, kg) | Change from baseline visit to final 3-month period
  Average baseline and final visit (Muscle Mass MM, kg)

OTHER OUTCOMES:
Treatment-related adverse events | Change from baseline visit to final 3 months
  Presence of adverse events, suspected adverse reactions and adverse reactions to treatment, on a scale of:
  A) Mild. They present with easily tolerated signs and symptoms, do not require treatment, do not prolong hospitalization and may or may not require discontinuation of the medication.
  B) Moderate. They interfere with normal activities (and may cause absences from work or school), without directly threatening the patient's life. They require pharmacological treatment and may or may not require discontinuation of the medication causing the adverse reaction.
  C) Severe. They interfere with normal activities (and may cause absences from work or school), directly threaten the patient's life. They require pharmacological treatment and require discontinuation of the medication causing the adverse reaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No